CLINICAL TRIAL: NCT01505686
Title: MRI Findings in Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, Principal investigator, North Karelia Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NKCH-Surg-008
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Inguinal Hernia; Pain
MeSH Terms: conditions — Hernia, Inguinal; Pain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group (Experimental): All patients in this study have MRI scan prior to hernia repair surgery. If inflammatory changes are present, the scan is repeated 6 months after surgery. If not, the scan is performed only if the patient has pain problems at 6 months.
  Interventions: Procedure: MRI scan

INTERVENTIONS:
Procedure: MRI scan — MRI scan with a 1,5 T MRI scanner

SUMMARY:
MRI imaging in clinically evident inguinal hernia is not routinely used. In other painful inguinal conditions (such as sportsmans hernia) inflammatory changes have been detected. The aim of the present study is to determine, whether similar inflammatory changes can be detected with MRI scan in inguinal hernia. Also, patient questionaires are used preoperatively and postoperatively to determine, if preoperative pain scores can be used as a predictive value for postoperative prolonged pain/neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* age < 50 years
* painful inguinal hernia

Exclusion Criteria:

* conditions that do not allow the use of MRI
* conditions that prevent general anesthesia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory changes in MRI scan | 7 months
  MRI scan is performed preoperatively and 6 months postoperatively to find possible inflammatory changes in the inguinal area, and the changes that a hernia mesh repair causes. If preoperative MRI scan does not have inflammatory changes, 6-month-MRI is only performed on-demand (if the patient is experiencing prolonged pain.

SECONDARY OUTCOMES:
Pain scores | 7 months
  Preoperative and postoperative patient questionaires are used. Preoperative values are examined to determine, if they can be used to predict postoperative pain problems.

CONTACTS AND LOCATIONS:
Locations (1):
- North Karelia Central Hospital, department of surgery, Joensuu, Finland